CLINICAL TRIAL: NCT06679764
Title: Comparison Between the Ultrasound Guided Pericapsular Nerve Group Block and Anterior Quadratus Lumborum Block in Elderly Patients Undergoing Total Hip Replacement Surgeries: A Randomized Controlled Clinical Trial
Brief Title: The Ultrasound Guided Pericapsular Nerve Group and Anterior Quadratus Lumborum Blocks in Hip Replacement Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Youssef, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MD-16-2022
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Post Operative Analgesia
MeSH Terms: interventions — Dental Occlusion; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Anterior quadratus lumborum block technique (AQLB) (Active Comparator): AQLB performed in the lateral position. A low-frequency convex probe for the abdomen (2-5) MHz convex probe, (Siemens ACUSON X300 Ultrasound System) was placed horizontally above the iliac crest. On ultrasound, The psoas major was located on the ventral side of the transverse process, the erector spinae was located on the dorsal side of the transverse process, and the quadratus lumborum was located on the lateral side of the transverse process.
  A 38-mm 22-gauge regional block needle was advanced in-plane from posterior to anterior directing the needle tip in the fascial plane between the psoas major and the quadratus lumborum that was confirmed by injecting 1 ml saline and watchingt the fluil fting the muscle while not distending any of the two muscles (hydro-localization). Then 30mL of local anaesthetic (29ml of 0.25% bupivacaine + 1 ml of dexamethasone (4mgs) was injected with observation of local anaesthesia spread in the fascial plane.
  Interventions: Procedure: Anterior quadratus lumborum block technique (AQLB)
- Pericapsular Nerve Group (PENG) block (Active Comparator): With the patients in supine position, A low-frequency convex probe (2-5 MHz) in was placed in a transverse plane over the anterior inferior iliac spine and then it was rotated 45 degrees in counter-clockwise direction to be aligned with the pubic ramus. In this view, the ilio-pubic eminence, iliopsoas muscle tendon, femoral nerve and vessels was observed. With in-plane approach, a 38-mm 22-gauge (22-G, 50-mm) regional block needle inserted in-plane, from lateral to medial to place the needle tip underneath the iliopsoas tendon, exactly between the ilipsoas fascia anteriorly and the pubic ramus posteriorly. Following negative resistance and aspiration tests, correct location of the needle tip was confirmed by injecting 1 ml saline. Then, 30mL of local anaesthetic (29ml of 0.25% bupivacaine+ 1ml of dexamethasone (4mgs) was injected while observing for adequate fluid spread.
  Interventions: Procedure: Pericapsular Nerve Group (PENG) block
- Control Group (Active Comparator): Pataints received opioid analgesia with GA
  Interventions: Drug: Control Group

INTERVENTIONS:
Procedure: Anterior quadratus lumborum block technique (AQLB) — AQLB performed in the lateral position. A low-frequency convex probe for the abdomen (2-5) MHz convex probe, (Siemens ACUSON X300 Ultrasound System) was placed horizontally above the iliac crest. On ultrasound, The psoas major was located on the ventral side of the transverse process, the erector spinae was located on the dorsal side of the transverse process, and the quadratus lumborum was located on the lateral side of the transverse process.
  A 38-mm 22-gauge regional block needle was advanced in-plane from posterior to anterior directing the needle tip in the fascial plane between the psoas major and the quadratus lumborum that was confirmed by injecting 1 ml saline and watchingt the fluil fting the muscle while not distending any of the two muscles (hydro-localization). Then 30mL of local anaesthetic (29ml of 0.25% bupivacaine + 1 ml of dexamethasone (4mgs) was injected with observation of local anaesthesia spread in the fascial plane.
  Arms: Anterior quadratus lumborum block technique (AQLB)
Procedure: Pericapsular Nerve Group (PENG) block — With the patients in supine position, A low-frequency convex probe (2-5 MHz) in was placed in a transverse plane over the anterior inferior iliac spine and then it was rotated 45 degrees in counter-clockwise direction to be aligned with the pubic ramus. In this view, the ilio-pubic eminence, iliopsoas muscle tendon, femoral nerve and vessels was observed. With in-plane approach, a 38-mm 22-gauge (22-G, 50-mm) regional block needle inserted in-plane, from lateral to medial to place the needle tip underneath the iliopsoas tendon, exactly between the ilipsoas fascia anteriorly and the pubic ramus posteriorly. Following negative resistance and aspiration tests, correct location of the needle tip was confirmed by injecting 1 ml saline. Then, 30mL of local anaesthetic (29ml of 0.25% bupivacaine+ 1ml of dexamethasone (4mgs) was injected while observing for adequate fluid spread.
  Arms: Pericapsular Nerve Group (PENG) block
Drug: Control Group — Pataints received opioid analgesia with genaral anesthesia
  Arms: Control Group

SUMMARY:
The investigators hypothesis that PENG block will produce effective opioid sparing analgesia with enhanced motor recovery more than AQLB in elderly patients undergoing total hip replacement surgeries

DETAILED DESCRIPTION:
Aim of the work:

The aim of this study is to compare analgesic efficacy and motor recovery of the ultrasound guided anterior quadratus lumborum block and the pericapsular nerve group block

Statistical Analysis:

Data will be coded and entered using the statistical package SPSS version 22. Categorical data will be expressed frequency and proportion and will be compared by Chi2. Numerical data will be summarized using mean and standard deviation. Comparisons between groups for normally distributed data will be done using analysis of variance (ANOVA), while for non-normally distributed numeric variable will be done by Krauskal Wallis test. P value less than or equal to 0.05 will be considered statistically significant. All test will be two tailed

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Type of surgery; unilateral elective total hip replacement.
* Physical status ASA I- III
* Age ≥ 65 Years.
* Body mass index (BMI): > 20 kg/m2 and < 35 kg/m2.
* Traumatic fracture hip through anterolateral approach.

Exclusion Criteria:

* Patient refusal.
* Patients with known sensitivity or contraindication to drugs used in the study (local anesthetics & opioids).
* History of psychological disorders and/or chronic pain.
* Pre- existing peripheral neuropathies
* Coagulopathy.
* Infection of the skin at the site of needle puncture area.
* Active cardiac condition (unstable coronary syndromes, significant arrhythmias, severe valvular disease).
* Acute respiratory disease (active chest infection, respiratory failure).
* Advanced liver disease (increased liver enzymes >3 folds) or severe kidney disease (creatinine >2).
* long operative time more than 3 hours.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Ollaek, MD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Egypt

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Elderly patients (≥65 years) with traumatic hip fractures scheduled for elective unilateral total hip arthroplasty via an anterolateral approach under general anesthesia were recruited at the Orthopedic Surgical Theater, Cairo University Hospital. Recruitment occurred at a single tertiary university hospital in Egypt.
Pre-assignment Details: No wash-out or run-in phase. All eligible, consenting patients were randomized 1:1:1 immediately before surgery after induction of general anesthesia. No participants were excluded after enrollment and before assignment to study arms.
Groups:
- Anterior Quadratus Lumborum Block Technique (AQLB): Single-shot ultrasound-guided anterior quadratus lumborum block performed after induction of GA. 30 mL local anesthetic mixture (29 mL 0.25% bupivacaine + 1 mL dexamethasone 4 mg) injected in the fascial plane between quadratus lumborum and psoas major muscles using an in-plane posterior-to-anterior approach.
- Pericapsular Nerve Group (PENG) Block: Single-shot ultrasound-guided pericapsular nerve group (PENG) block performed after induction of GA. 30 mL local anesthetic mixture (29 mL 0.25% bupivacaine + 1 mL dexamethasone 4 mg) injected in the fascial plane between iliopsoas tendon and superior pubic ramus under ultrasound guidance.
- Control Group: General anesthesia without regional block. Intraoperative fentanyl administered as required; post-operative IV morphine (0.05 mg/kg boluses, maximum 0.3 mg/kg/24 h) as rescue analgesia within a multimodal regimen including IV paracetamol.
Period: Overall Study
Arm/Group | Anterior Quadratus Lumborum Block Technique (AQLB) | Pericapsular Nerve Group (PENG) Block | Control Group
Started | 31 | 31 | 31
Completed | 31 | 31 | 31
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were obtained for all randomized participants in each arm (31 per group), with no exclusions.
Groups:
- Total: Total of all reporting groups
Arm/Group | Anterior Quadratus Lumborum Block Technique (AQLB) | Pericapsular Nerve Group (PENG) Block | Control Group | Total
Number analyzed (Participants) | 31 | 31 | 31 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 31 | 31 | 31 | 93
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 12 | 47
  Male | 14 | 13 | 19 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Egypt | 31 | 31 | 31 | 93
Age [Median (Standard Deviation); unit: years] | 68.74 (3.32) | 70.87 (4.74) | 69.55 (2.59) | 69.72 (3.73)

OUTCOME MEASURES:

1. Primary Outcome: The Total Amount of Morphine Consumption
Description: Total dose of IV morphine (mg) administered as rescue analgesia during the first 24 postoperative hours. Morphine 0.05 mg/kg IV boluses were given when NRS ≥4, up to a maximum of 0.3 mg/kg/24 h. Reported as median (IQR).
Time Frame: Immediatly post operative for 24 hours
Population: All randomized participants (N=93; 31 per group) received the allocated intervention and completed 24-hour follow-up; no losses to follow-up and no exclusions from analysis. Primary outcome data were available for all participants; analysis was performed on the full randomized set (intention-to-treat).
Measure: Median (Inter-Quartile Range); unit: mg of IV morphine
Arm/Group | Anterior Quadratus Lumborum Block Technique (AQLB) | Pericapsular Nerve Group (PENG) Block | Control Group
Number analyzed (Participants) | 31 | 31 | 31
mg of IV morphine | 6.0 [3.5 to 8.0] | 8.0 [6.0 to 11.0] | 12.0 [10.5 to 12.0]
Statistical Analysis 1: Comparison: Anterior Quadratus Lumborum Block Technique (AQLB) vs Pericapsular Nerve Group (PENG) Block vs Control Group; Comparison of total 24-h postoperative morphine consumption across three groups using Kruskal-Wallis test; post-hoc pairwise Mann-Whitney tests with Bonferroni correction; Test type: Superiority — Non-parametric analysis due to non-normal distribution. AQLB < PENG < Control for median morphine use. Significant pairwise differences: PENG vs Control, AQLB vs Control, and PENG vs AQLB (P=0.035); p = 0.035, Kruskal-Wallis — Overall comparison of 24-h postoperative morphine consumption across the three groups used the Kruskal-Wallis test (non-parametric)

2. Secondary Outcome: Numeric Pain Rating Scale at Rest Over First 24 Hours
Description: Pain intensity at rest using 0-10 Numeric Pain Rating Scale (0 = no pain, 10 = worst imaginable pain) measured at specified time points; data reported as median (IQR).
Time Frame: 30 minutes, 2, 4, 6, 8, 12, 18, and 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Anterior Quadratus Lumborum Block Technique (AQLB) | Pericapsular Nerve Group (PENG) Block | Control Group
Number analyzed (Participants) | 31 | 31 | 31
units on a scale
  30 min | 0.0 [0.0 to 0.0] | 1.0 [0.0 to 1.0] | 2.0 [2.0 to 3.0]
  2 h | 1.0 [0.0 to 1.0] | 1.0 [0.0 to 1.0] | 2.0 [1.0 to 6.0]
  4 h | 1.0 [1.0 to 2.0] | 2.0 [0.0 to 2.0] | 3.0 [2.0 to 3.0]
  6 h | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  8 h | 2.0 [2.0 to 3.0] | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0]
  12 h | 3.0 [2.0 to 3.0] | 3.0 [3.0 to 4.0] | 3.0 [2.0 to 3.0]
  18 h | 3.0 [2.0 to 3.0] | 3.0 [3.0 to 4.0] | 3.0 [2.0 to 4.0]
  24 h | 3.0 [3.0 to 3.0] | 3.0 [3.0 to 4.0] | 3.0 [2.0 to 3.0]

3. Secondary Outcome: Numeric Pain Rating Scale During Passive 90° Hip Flexion Over First 24 Hours
Description: Pain intensity during passive 90° hip flexion using 0-10 NRS at same time points; reported as median (IQR).
Time Frame: at 30 minutes, 2, 4, 6, 8, 12, 18 and 24 hours postoperatively
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Anterior Quadratus Lumborum Block Technique (AQLB) | Pericapsular Nerve Group (PENG) Block | Control Group
Number analyzed (Participants) | 31 | 31 | 31
units on a scale
  30 min | 1.0 [1.0 to 1.0] | 1.0 [0.0 to 2.0] | 3.0 [3.0 to 3.0]
  2 h | 2.0 [1.0 to 2.0] | 1.0 [0.0 to 2.0] | 5.0 [3.0 to 7.0]
  4 h | 2.0 [2.0 to 3.0] | 2.0 [1.0 to 3.0] | 3.0 [3.0 to 4.0]
  6 h | 3.0 [2.0 to 3.0] | 3.0 [1.0 to 3.0] | 3.0 [3.0 to 7.0]
  8 h | 3.0 [3.0 to 3.0] | 3.0 [2.0 to 4.0] | 5.0 [3.0 to 6.0]
  12 h | 3.0 [3.0 to 4.0] | 3.0 [3.0 to 4.0] | 3.0 [3.0 to 3.0]
  18 h | 3.0 [3.0 to 4.0] | 4.0 [3.0 to 5.0] | 5.0 [4.0 to 7.0]
  24 h | 3.0 [3.0 to 4.0] | 3.0 [3.0 to 4.0] | 3.0 [3.0 to 4.0]

4. Secondary Outcome: Time to First Rescue Morphine Analgesia
Description: Time from arrival in PACU to first administration of IV morphine rescue dose (NRS ≥4). Reported as median (IQR).
Time Frame: Immediatly post operative for 24 hours
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Anterior Quadratus Lumborum Block Technique (AQLB) | Pericapsular Nerve Group (PENG) Block | Control Group
Number analyzed (Participants) | 31 | 31 | 31
Hours | 12.0 [6.0 to 18.0] | 8.0 [7.0 to 12.0] | 2.0 [2.0 to 4.0]

5. Secondary Outcome: Manual Muscle Test (MMT) Score for Quadriceps/Iliopsoas Over First 24 Hours
Description: Manual muscle test (0-5 scale; 0 = no contraction, 5 = full ROM against gravity and maximal resistance) for quadriceps and iliopsoas muscles on the operated side, after extubation, at predefined time points.
Time Frame: 30 minutes, 2, 4, 6, 8, 12, 18 and 24 hours postoperatively
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Anterior Quadratus Lumborum Block Technique (AQLB) | Pericapsular Nerve Group (PENG) Block | Control Group
Number analyzed (Participants) | 31 | 31 | 31
units on a scale
  30 min | 1.0 [0.0 to 1.0] | 2.0 [2.0 to 2.0] | 0.0 [0.0 to 2.0]
  2 h | 1.0 [1.0 to 1.0] | 3.0 [3.0 to 3.0] | 1.0 [1.0 to 1.0]
  4 h | 2.0 [2.0 to 2.0] | 3.0 [3.0 to 4.0] | 2.0 [2.0 to 3.0]
  6 h | 2.0 [2.0 to 3.0] | 4.0 [4.0 to 4.0] | 3.0 [2.0 to 4.0]
  8 h | 3.0 [3.0 to 3.0] | 4.0 [4.0 to 4.0] | 3.0 [3.0 to 4.0]
  12 h | 3.0 [3.0 to 3.0] | 4.0 [4.0 to 4.0] | 4.0 [3.0 to 4.0]
  18 h | 3.0 [3.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  24 h | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]

6. Secondary Outcome: Active Hip Flexion Range of Motion (0°-90°) Over First 24 Hours
Description: Active hip flexion range of motion (degrees) of the operated hip, from 0° to 90°, assessed at same time points as MMTe. Reported as median (IQR).
Time Frame: 30 minutes, 2, 4, 6, 8, 12, 18 and 24 hours postoperatively
Measure: Median (Inter-Quartile Range); unit: Degrees of hip flexion
Arm/Group | Anterior Quadratus Lumborum Block Technique (AQLB) | Pericapsular Nerve Group (PENG) Block | Control Group
Number analyzed (Participants) | 31 | 31 | 31
Degrees of hip flexion
  30 min | 0.0 [0.0 to 0.0] | 20.0 [10.0 to 20.0] | 0.0 [0.0 to 10.0]
  2 h | 0.0 [0.0 to 0.0] | 30.0 [20.0 to 45.0] | 20.0 [0.0 to 20.0]
  4 h | 0.0 [0.0 to 20.0] | 45.0 [30.0 to 45.0] | 30.0 [20.0 to 45.0]
  6 h | 0.0 [0.0 to 20.0] | 45.0 [45.0 to 45.0] | 45.0 [30.0 to 45.0]
  8 h | 30.0 [20.0 to 45.0] | 90.0 [45.0 to 90.0] | 45.0 [30.0 to 45.0]
  12 h | 45.0 [45.0 to 45.0] | 90.0 [90.0 to 90.0] | 45.0 [45.0 to 60.0]
  18 h | 45.0 [45.0 to 45.0] | 90.0 [90.0 to 90.0] | 45.0 [45.0 to 60.0]
  24 h | 90.0 [45.0 to 90.0] | 90.0 [90.0 to 90.0] | 45.0 [45.0 to 90.0]

7. Secondary Outcome: Total Intraoperative Fentanyl Dose
Description: Total dose of IV fentanyl administered intraoperatively. Additional boluses of 1 μg/kg were given if MAP or HR increased by >20% above baseline. Reported as mean ± SD.
Time Frame: During surgery
Measure: Mean (Standard Deviation); unit: μg fentanyl
Arm/Group | Anterior Quadratus Lumborum Block Technique (AQLB) | Pericapsular Nerve Group (PENG) Block | Control Group
Number analyzed (Participants) | 31 | 31 | 31
μg fentanyl | 142.58 (18.43) | 152.90 (60.23) | 236.61 (90.68)

8. Secondary Outcome: Time to First Walk
Description: Time from end of surgery to first ambulation (≥3 steps with walker). Reported as median (IQR)
Time Frame: From end of surgery until first walk (within postoperative 24 h)
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Anterior Quadratus Lumborum Block Technique (AQLB) | Pericapsular Nerve Group (PENG) Block | Control Group
Number analyzed (Participants) | 31 | 31 | 31
Hours | 24.0 [18.0 to 24.0] | 8.0 [8.0 to 12.0] | 18.0 [12.0 to 24.0]

9. Secondary Outcome: Length of Hospital Stay
Description: Time from surgery to hospital discharge. Reported as mean ± SD.
Time Frame: From date of surgery until discharge
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Anterior Quadratus Lumborum Block Technique (AQLB) | Pericapsular Nerve Group (PENG) Block | Control Group
Number analyzed (Participants) | 31 | 31 | 31
Days | 3.16 (0.52) | 2.13 (0.34) | 2.94 (0.68)

ADVERSE EVENTS:
Time Frame: Intraoperative period and first 24 postoperative hours through discharge up to 4 days
Description: Adverse events were prospectively monitored intraoperatively and during the first 24 h postoperatively. Predefined events included block-related complications (sedation, hallucination, respiratory depression, hematoma, lower limb weakness, hypotension, falls) and morphine-related postoperative nausea and vomiting (PONV).
Arm/Group | Anterior Quadratus Lumborum Block Technique (AQLB) | Pericapsular Nerve Group (PENG) Block | Control Group
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 7/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anterior Quadratus Lumborum Block Technique (AQLB) (N=31) | Pericapsular Nerve Group (PENG) Block (N=31) | Control Group (N=31)
Postoperative nausea and vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 7 (7)

LIMITATIONS AND CAVEATS:
Single-center study at a tertiary university hospital, which may limit generalizability. Pain and motor assessments are partly subjective. Follow-up was restricted to the first 24 postoperative hours; long-term functional outcomes and block-related complications beyond this period were not assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT06679764/Prot_SAP_000.pdf